CLINICAL TRIAL: NCT01305473
Title: A Single Arm, Single-Center, Retrospective Study With Prospective Follow-Up of Laparoscopic Ventral Hernia Repair Utilizing the Bard Sepramesh IP Composite
Brief Title: A Retrospective Study With Prospective Follow-Up of Laparoscopic Ventral Hernia Repair Utilizing the Bard Sepramesh IP Composite
Acronym: Sepramesh
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: DVL-HE007
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sepramesh Group

SUMMARY:
This study will enroll subjects who underwent a laparoscopic ventral hernia repair utilizing Sepramesh at least 12 months before starting in this study.

The consented subjects' medical records will be reviewed for evidence of any risk factors of hernia recurrence, procedure time, complications and any documented recurrences. The subjects will be asked to undergo a physical exam to rule out any recurrences that were not documented in the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone a laparoscopic ventral repair utilizing Sepramesh at least 12 months before starting in this study.
* Have signed an Informed Consent Form (ICF).

Exclusion Criteria:

* Underwent implantation of Sepramesh for any reason other than ventral hernia repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been treated with Sepramesh at least 12 months before starting in this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Archer, MD, Principal Investigator — Providence Medical Group and Cornerstone Medical Center
Locations (1):
- Cornerstone Medical Center, Centerville, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2010 and February 2011, a total of 90 subjects were enrolled at a single study site.
Groups:
- Sepramesh Group: Subjects who underwent laparoscopic ventral hernia repair utilizing Bard Sepramesh Composite at least 12 months prior to enrollment.
Period: Overall Study
Arm/Group | Sepramesh Group
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 56.0 (12.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 87
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 90
Weight [Mean (Standard Deviation); unit: kilograms] | 98.5 (23.92)
Height [Mean (Standard Deviation); unit: centimeters] | 170.3 (10.16)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 33.9 (7.36)
Hernia Classification [Number; unit: participants] — Type of hernia subject had repaired during the index procedure: umbilical, incisional, or umbilical and incisional.
  participants
    Umbilical | 43
    Incisional | 42
    Umbilical and Incisional | 5

OUTCOME MEASURES:

1. Primary Outcome: Hernia Recurrence Rate of Hernias Post Repair With Sepramesh.
Description: A recurrent hernia is a hernia, confirmed by the Investigator at any point after the surgery, in the same location as the hernia repaired in the index procedure.
Time Frame: 12 months or greater (average follow-up time of 3 years; range 13-65 months)
Population: All enrolled subjects were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 90
participants | 1

2. Secondary Outcome: Complications in Subjects With Hernias Repaired With Sepramesh.
Description: Complications will be assessed by evaluation of the procedural and device related adverse events (AEs) documented in the subject's medical files from the time surgery was initiated until the day the subject had a postoperative visit (that is, the protocol specified postoperative visit for conducting a physical examination).
Time Frame: 12 months or greater (average follow-up time of 3 years; range 13-65 months)
Population: All enrolled subjects were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 90
participants | 2

3. Secondary Outcome: Procedural Time for Sepramesh Placement.
Description: Procedure time will be defined as beginning when the Investigator made the initial incision and ending when the skin closure was completed (skin to skin).
Time Frame: Day 0
Population: All enrolled subjects were included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 90
minutes | 41.4 (20.56)

4. Secondary Outcome: Recovery Time Associated With Hernias Repaired With Sepramesh.
Description: Recovery time will be defined as the time it took for the subject to return to work.
Time Frame: 12 months or greater (average follow-up time of 3 years; range 13-65 months)
Population: Data not available: none of the subject medical records reported return to work data. Secondary endpoint analysis could not be performed.
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 0

5. Post Hoc Outcome: Hernia Recurrence Rate of Incisional Hernias Post Repair With Sepramesh.
Description: A recurrent incisional hernia is an incisional hernia, confirmed by the Investigator at any point after the surgery, in the same location as the incisional hernia that was repaired in the index procedure.
Time Frame: 12 months or greater
Population: The analysis population included the 42 subjects who underwent surgery to repair incisional hernias in the index procedure.
Measure: Number; unit: participants
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 42
participants | 1

6. Post Hoc Outcome: Hernia Recurrence Rate of Umbilical Hernias Post Repair With Sepramesh.
Description: A recurrent umbilical hernia is an umbilical hernia, confirmed by the Investigator at any point after the surgery, in the same location as the umbilical hernia that was repaired in the index procedure.
Time Frame: 12 months or greater
Population: The analysis population included the 43 subjects who underwent surgery to repair umbilical hernias in the index procedure.
Measure: Number; unit: participants
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 43
participants | 0

7. Post Hoc Outcome: Hernia Recurrence Rate Post Repair With Sepramesh in Subjects With Both Incisional and Umbilical Hernias
Description: A recurrent hernia is a hernia (either umbilical or incisional), confirmed by the Investigator at any point after surgery, in the same location as the hernia repaired in the index procedure.
Time Frame: 12 months or greater
Population: This analysis included the 5 subjects who underwent surgery to repair both incisional and umbilical hernias in the index procedure.
Measure: Number; unit: participants
Arm/Group | Sepramesh Group
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Time Frame: Protocol defined adverse events were collected for a period of 12 months or greater, with the collection period beginning at the time of the index procedure and ending at the time of the subject's last study contact.
Description: Adverse events (or complications) were defined as any undesirable clinical event occurring in the abdominal skin, abdominal wall, involving abdominal organs and/or any other event judged to be related to the surgical procedure of Sepramesh Composite.
Arm/Group | Sepramesh Group
Serious Adverse Events (participants affected / at risk) | 3/90
Other Adverse Events (participants affected / at risk) | 1/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sepramesh Group (N=90)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) — This event is the hernia recurrence identified in the primary outcome analysis. It was reported approximately 14 months after the hernia repair procedure. Event was reported as serious but mild and possibly related to the hernia repair procedure.
Seroma (Injury, poisoning and procedural complications) | 1 (1) — Postoperative seroma reported following a procedure which was unrelated to both the study device or procedure. Event was reported as serious but mild and unrelated to both the device and the procedure.
Postoperative hernia (Injury, poisoning and procedural complications) | 1 (1) — Subject developed a new (non-study) hernia at an instrument insertion site used during the procedure to repair the study hernia. Event was reported as serious but mild, unrelated to the device and definitely related to the procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sepramesh Group (N=90)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was designed to use existing data. Limitations include: limited data generalizability given the retrospective, single center study design; incomplete documentation did not permit evaluation of recovery time as pre-specified secondary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days